CLINICAL TRIAL: NCT05309603
Title: Alterations in Gait, Strength, and Power After Ruck Marching
Acronym: SPARTAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Assistant Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00006175
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Exercise; Fatigue
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unloaded Walking (Active Comparator): Walking on a treadmill without wearing a pack
  Interventions: Other: Walking
- Loaded Walking High (Experimental): Walking on a treadmill while wearing a 30% body mass load with the weight placed at the high-back
  Interventions: Other: Loaded Walking High
- Loaded Walking Mid (Experimental): Walking on a treadmill while wearing a 30% body mass load with the weight placed at the mid-back
  Interventions: Other: Loaded Walking Mid

INTERVENTIONS:
Other: Loaded Walking High — Walking three miles on a treadmill at a self-selected speed while wearing a backpack with weight carried high on the back
  Arms: Loaded Walking High
Other: Loaded Walking Mid — Walking three miles on a treadmill at a self-selected speed while wearing a backpack with weight carried on the mid-back
  Arms: Loaded Walking Mid
Other: Walking — Walking three miles on a treadmill at a self-selected speed
  Arms: Unloaded Walking

SUMMARY:
The purpose of this study is to determine change in injury risk and performance variables in males and females after walking unloaded and carrying a load with two different distributions (high-pack placement and mid-pack placement) to identify differences in injury risk

ELIGIBILITY:
Inclusion Criteria:

* Healthy, physically active individuals
* 18-39 years old

Exclusion Criteria:

* History of musculoskeletal injury within the last six months or still under a physicians care for an injury occurring more than six month prior
* History of spinal disc injury
* History of cardiovascular, metabolic, respiratory, neural, or renal disease
* No previous history or education of completing resistance exercise
* Hypertensive or tachycardic during the screening visit (SBP > 139 mmHg, DBP > 89 mmHg, heart rate > 100 bpm)
* Taking medication or supplements with a known side effect of affecting physiologic responses to exercise (e.g., beta blockers, omega-3 fatty acids, statins, aspirin)
* Any form of tobacco or nicotine use
* A positive pregnancy test at any point in the study
* Study physician discretion based on any other medical condition or medication
* Gastrointestinal disease or previous surgery prohibiting internal body temperature pill use. Subjects who have any contraindication to internal body temperature pill ingestion will be given the option to insert the pill rectally (as a suppository) or use a rectal probe.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen Consumption | Upon completion of 3 miles of walking, an average of 45 minutes
  Oxygen consumption will be measured using indirect calorimetry
Increased muscular jerk | Upon completion of 3 miles of walking, an average of 45 minutes
  Jerk will be measured using accelerometers placed at the torso and ankle

CONTACTS AND LOCATIONS:
Overall Officials: Riana Pryor, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers.